CLINICAL TRIAL: NCT00206895
Title: Photodynamic Therapy of Acne Vulgaris - a Randomized Blinded Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KF-01-177/04
Record Dates: First submitted 2005-09-12; First posted 2005-09-21 (Estimated); Last update posted 2006-10-11 (Estimated); Status verified 2004-10

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Photochemotherapy

INTERVENTIONS:
Procedure: Photodynamic therapy

SUMMARY:
The purpose of the study is to evaluated the efficacy and tolerability of methyl aminolevulinate and 5-aminolevulinic acid photodynamic therapy in patients with moderate to severe facial acne vulgaris in a randomized controlled and investigator blinded trial.

ELIGIBILITY:
Inclusion Criteria:18 years or older, good health, more than 12 inflammatory facial acne lesions -

Exclusion Criteria:skin type VI, pregnant or lactating woman. Oral retinoid use within one year, systemic antibiotics within 1 month, topical acne treatment within 2 weeks.

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2004-11

PRIMARY OUTCOMES:
Lesion counts (non-inflammatory and inflammatory)
Leeds Revised Acne Grading System

SECONDARY OUTCOMES:
Pain
Side effects

CONTACTS AND LOCATIONS:
Overall Officials: Hans Christian Wulf, MD, Sci, Study Director — Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen, Copenhagen NV, Denmark